CLINICAL TRIAL: NCT06478342
Title: Left Atrial Function After Pulsed Field Ablation of Atrial Fibrillation
Status: Not yet recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Marek Hozman, electrophysiologist, Charles University, Czech Republic
Other Study IDs: PFA - strain
Record Dates: First submitted 2024-06-22; First posted 2024-06-27 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; pulsed field ablation; left atrial strain
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Prospective cohort: Non-paroxysmal AF patients
  Interventions: Procedure: ablation

INTERVENTIONS:
Procedure: ablation — Pulsed field ablation, MRI and TEE examinations (LA strain)

SUMMARY:
Introduction: Pulsed field ablation (PFA) has emerged in routine clinical practice as a new promising technology in catheter-based treatment of atrial fibrillation (AF). The ease of PFA technology enables more extensive ablation in shorter time. On one hand, extensive ablation is advocated to decrease the AF recurrence in persistent patients, on the other hand it is an important predictor of developing left atrial stiff syndrome with a reported incidence rate of 3.7 - 8.2 % in persistent patients during the era of radiofrequency ablation.

Goals of the study: The main hypothesis is that the LA function (strain) will tend to decline after extensive PFA. It will be assessed using transthoracic echocardiography (TTE) and magnetic resonance (MRI).

Secondary endpoint analysis will include the evaluation of the distribution of late gadolinium enhancement (LGE) after ablation compared to baseline scans, evaluation of heart failure biomarkers after ablation, and description of the rate of AF recurrence.

Methods: This project is a prospective, nonrandomised, two-centre (University Hospital Kralovske Vinohrady and University Hospital Motol) observational study including 50 non-paroxysmal AF patients with indication for catheter ablation. Before the ablation, all patients will undergo LGE MRI and TTE (after cardioversion if AF present). The ablation procedure will be performed using pulsed field technology and will include pulmonary vein isolation, posterior wall ablation and mitral isthmus ablation. Patients will be followed for 6 months. 3 months after the ablation, LGE MRI will be performed. TTE examinations will be carried out on the day after the ablation, at 3 and at 6 months. Heart failure biomarkers (N-terminal proatrial natriuretic peptide, fibroblast growth factor 23, and galectin 3) levels will be analysed at baseline, and 3 and 6 months after the procedure. ECG Holter monitoring will be performed at 3- and 6-months visits.

ELIGIBILITY:
Inclusion Criteria:

* Non-paroxysmal AF with an indication for catheter ablation
* Age above 18
* Signed informed consent

Exclusion Criteria:

* Contraindication to MRI
* BMI > 35 kg/m2
* Contraindication to amiodarone
* Left atrial size > 60 mm
* History of any LA ablation
* Significant valvular disease (mitral regurgitation ¾ or greater, moderate or severe aortic stenosis)
* Severe pulmonary hypertension
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for AF ablation procedures
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Changes in LA function (strain) by MRI (baseline vs. 3m values) | Baseline MRI to 3 months after procedure
  LA strain (baseline vs. 3 months)
Changes in LA function (strain) by TTE (baseline vs. 3m values) | Procedure to 3 months
  LA strain (baseline vs. 3 months)

SECONDARY OUTCOMES:
Changes in LA fibrosis distribution (LGE MRI) (baseline vs. 3 m values) | Baseline MRI to 3 months after procedure
  LGE evaluation (baseline vs. 3 months MRI)
Changes in ANP, FGF 23, GAL 3 levels (baseline vs. 3 m values) | baseline vs. 3 m values
  laboratory analysis
AF freedom | Procedure to 6 months visit
  defined as an absence of AF/atrial tachycardia lasting > 30 s during follow-up including Holter monitoring
Changes in strain function on TTE over time | baseline TTE to 6 months control
  comparison of strain values obtained at all 4 time points

IPD SHARING:
Plan to Share IPD: No